CLINICAL TRIAL: NCT02461784
Title: The Effect of Methotrexate on Sperm Quality in Men With Inflammatory Bowel Disease
Status: Terminated | Type: Observational
Why Stopped: slow enrollment per COVID-19 pandemic and staffing resources
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0487; MTX/Sperm in IBD (Other: UW-Madison Study Staff); Protocol Version 8/24/2015 (Other: UW Madison); A534250 (Other: UW Madison); SMPH\MEDICINE\GASTROENT (Other: UW Madison)
Record Dates: First submitted 2015-05-26; First posted 2015-06-03 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2022-09

CONDITIONS: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Seeds; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Male subjects with IBD diagnosis currently taking methotrexate (MTX) as treatment for their disease.
  Interventions: Procedure: Semen & Data Collection
- Control: Male subjects with IBD diagnosis not exposed to methotrexate (MTX) as treatment for their disease.
  Interventions: Procedure: Semen & Data Collection

INTERVENTIONS:
Procedure: Semen & Data Collection — If participants decide to participate in this research they will be asked to complete the informed consent process as well as asked a few questions such as age and race/ethnicity. If participants volunteered for this study because tehy have IBD, investigators will also collect some information from the participants medical record. Completing this portion of participation will take less than 1 hour.
  Participants will then be scheduled to complete the semen collection at the UW Health Generations Fertility Clinic located at 2365 Deming Way in Middleton, WI. This collection visit will take less than 1 hour to complete. Once participants have finished the collection visit they will have completed their participation in this research project.

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract which includes Crohn's disease (CD) and ulcerative colitis (UC) which peak in incidence (rate or frequency) during the reproductive years. An increasing number of young people will face challenging decisions regarding medical management of this chronic disease during a period of time when they are still completing schooling, establishing their career, and/or are building a family.

Treatment options for IBD consist of immunosuppressive therapy, such as immunomodulators (azathioprine and methotrexate). Methotrexate (MTX) is a folic acid antagonist (a substance that interferes with or inhibits the action of another). It is thought that MTX works by decreasing the inflammation in the gastrointestinal tract. MTX has been studied for many years and in used as treatment in not only IBD, but also in conditions such as rheumatoid arthritis and lupus. However, due to concerns about the safety of MTX, particularly in regards to fertility and pregnancy has limited its current use.

Participants are invited to take part in this research project to determine whether the treatment of IBD patients with MTX is associated with an increased risk for infertility. Investigators will recruit 75 male IBD patients under MTX treatment for their IBD as well as 75 healthy male controls for a total of 150 patients at the University of Wisconsin Hospital & Clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Cases: Men aged 18 to 40 years with a confirmed diagnosis of UC or CD based on endoscopy, pathology, and/or radiology AND who regularly take MTX (per oral, subcutaneous, or intramuscular) either as monotherapy or in combination with mesalamine (any except sulfasalazine), corticosteroids, anti-TNF agents, or anti-adhesion molecules for at least one month specifically for the treatment of IBD. Controls: Men aged 18 to 40 years with a confirmed diagnosis of UC or CD based on endoscopy, pathology, and/or radiology AND who do not take MTX (per oral, subcutaneous, or intramuscular) either as monotherapy or in combination with other IBD-specific drugs.
2. Individual able and willing to consent to donate their sperm to research.

Exclusion Criteria:

1. Men with previously documented problems with male reproductive health such as known hypothalamic-pituitary disorders (e.g. pituitary macroadenomas, pituitary infarction), primary hypogonadism (e.g. cryptorchidism, Klinefelter's syndrome), or disorders of sperm transport (e.g. erectile dysfunction, history of vasectomy)
2. Current use of alkylating agents, ketoconazole, sulfalsalazine, H2-receptor antagonists or spironolactone
3. Men who have undergone ileal pouch anal anastomosis within 3 months of study entry

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subject population will consist of individuals with inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Compare semen characteristics between male IBD patients on Methotrexate and non-methotrexate exposed males. | 12 month study
  The purpose of this study is to determine whether the treatment of IBD patients with MTX is associated with an increased risk for infertility using two different criteria for assessing male fertility: the WHO criteria for basic semen analysis and Fourier Harmonic Amplitudes. The latter will be used to describe nuclear shapes and sperm DNA staining intensity as this has been shown in animal models to correlate with male fertility. MTX-exposed male IBD patients (cases) will be compared with age-matched, non-MTX exposed patients (controls).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States